CLINICAL TRIAL: NCT02961335
Title: Validation of Alveolar Probe-based Confocal Laser Endomicroscopy Descriptors in Diffuse Parenchymal Lung Diseases : A Multicentric Prospective Study
Brief Title: Validation of Alveolar Probe-based Confocal Laser Endomicroscopy Descriptors in Diffuse Parenchymal Lung Diseases
Acronym: Microsemio-PI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/0208/HP
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Parenchymal Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Bronchoscopy; Chorionic Villi Sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient who need to undergo bronchoscopy (Experimental): Patient who need to undergo bronchoscopy. During bronchoscopy, biopsy sampling and Confocal microendoscopy will be done
  Interventions: Procedure: Bronchoscopy; Procedure: Confocal microendoscopy; Procedure: Biopsy sampling

INTERVENTIONS:
Procedure: Bronchoscopy — Patient who need to undergo bronchoscopy. During bronchoscopy, biopsy sampling and Confocal microendoscopy will be done
Procedure: Confocal microendoscopy — Confocal microendoscopy will be performed during this initial bronchoscopy
Procedure: Biopsy sampling — Patient who need to undergo bronchoscopy. During bronchoscopy, biopsy sampling and Confocal microendoscopy will be done

SUMMARY:
Diffuse parenchymal lung diseases (DPLD) include a variety of respiratory conditions that affect either the pulmonary interstitium or the alveolar space . The etiological diagnosis of DPLD is often challenging, because of the large number of pathological entities involved, which share close clinical and radiological presentations. High resolution Chest CT, a key diagnostic procedure in DPLD, is subject to significant inter-observer analysis variations, so that the diagnosis sometimes requires a surgical or transbronchial lung biopsy sampling. This invasive procedure is not devoid of morbidity and may be impossible to perform in fragile patients. Therefore, the definite diagnosis of DPLD is usually achieved following a multi-disciplinary expert consensus, based on careful medical history, chest CT and bronchoalveolar lavage examinations.

Alveolar probe-based confocal laser endomicroscopy (pCLE) is a mini invasive endoscopic technique that allows distal lung microscopic imaging in vivo, during a flexible bronchoscopy performed under topical anaesthesia. Since 2006, Alveolar pCLE has been used in a monocentric clinical trial at the Rouen University Hospital in more than 200 patients and healthy volunteers. This allowed the first pCLE in-vivo description of normal pulmonary acinus, and confirmed the safety of the technique.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* signed written informed consent
* indication for a flexible bronchoscopy
* DPLD characterized by clinical and radiological data compatible with : idiopathic pulmonary fibrosis (IPF), acute or chronic hypersensitivity pneumonitis (HPS), sarcoidosis, or asbestosis.
* Initial histological confirmation of the disease is not required for the inclusion of the patient and the realisation of the alveolar bronchoscopy.
* non-smoking or smoking cessation >6 month
* Patient affiliated with, or beneficiary of a social security category

Exclusion Criteria:

* respiratory failure and contraindication for a flexible bronchoscopy (this item will stay at the appreciation of the physician, arterial blood gaz sampling being not required)
* bleeding disorder which would be not compatible with the realization of a flexible bronchoscopy
* history of pneumonectomy or non functional lung controlateral to the pCLE procedure
* patients for which a per-endoscopic distal lung cryobiopsy is forecasted during the first diagnostic bronchoscopy,
* patients for which the bronchoscopy needs a general anesthesia and mechanical ventilation during the procedure
* anticoagulant or platelet aggregation inhibitors that cannot be interrupted for the flexible bronchoscopy
* patients for which a follow up or an adequate work-up to achieve the final diagnosis will not be possible.
* patients for which a cryobiopsy is forecasted during the bronchoscopy
* pregnant and breast feeding women, or women of childbearing potential not taking adequate contraception
* Patients unable to understand informed consent
* Patient on major legal measure of protection
* Patients participating in an other interventional clinical trial at the inclusion date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity of confocal imaging (solid pattern) for the diagnostic of the pulmonary nodule | Day 1
  Confocal imaging will be considered as "positive" when both
  * a solid pattern is displayed
  * a diagnostic biopsy is obtained at the site of confocal imaging

CONTACTS AND LOCATIONS:
Overall Officials: Luc THIBERVILLE, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No